CLINICAL TRIAL: NCT02072278
Title: Interventional, Randomised, Double-blind, Placebo-controlled, Active Comparator, Four-way Crossover Electroencephalography Study Investigating the Effects of Vortioxetine (Lu AA21004) in Healthy Male Subjects
Brief Title: Electroencephalography Study Investigating the Effects of Vortioxetine in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15835A; 2013-004015-53 (EudraCT Number)
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Men
MeSH Terms: interventions — Vortioxetine; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vortioxetine 10 mg (Experimental): encapsulated tablets; 3 daily doses in each treatment period; orally
  Interventions: Drug: Vortioxetine 10 mg
- Vortioxetine 20 mg (Experimental): encapsulated tablets; 3 daily doses in each treatment period; orally
  Interventions: Drug: Vortioxetine 20 mg
- Escitalopram 15 mg (Active Comparator): encapsulated tablets; 3 daily doses in each treatment period; orally
  Interventions: Drug: Escitalopram 15 mg
- Placebo (Placebo Comparator): capsules; 3 daily doses in each treatment period; orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine 10 mg
  Arms: Vortioxetine 10 mg
Drug: Vortioxetine 20 mg
  Arms: Vortioxetine 20 mg
Drug: Escitalopram 15 mg
  Arms: Escitalopram 15 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
To explore a neurophysiological marker (electroencephalography) of cognitive effect of vortioxetine

ELIGIBILITY:
Inclusion Criteria:

* The subject has a normal resting EEG at screening visit
* The subject is able to perform tasks with an auditory stimulus
* The subject is not visually impaired - normal prescription glasses are accepted
* The subject has a normal circadian rhythm, defined as a person who usually wakes between 6:00 and 9:00 a.m. and goes to sleep between 9:00 pm and midnight.

Exclusion Criteria:

* The subject has worked shifts, including night duty, or has travelled across >3 time zones <2 weeks prior to the first dose of IMP.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Battery of EEG measurements | The EEG task battery will be conducted on Days -1 and starting 6 hours post-dose on Days 1 and 3 of each treatment period.
  * Peak amplitude and latency of P300
  * AUC of qEEG power spectral bands delta, theta, alpha, beta and gamma
  * AUC of evoked gamma power spectral band
  * Peak amplitude and latency of N200
  * Peak amplitude and latency of error related negativity
  * Peak amplitudes and latencies in the evoked responses during successful versus non-successful encoding in the verbal memory task between treatments

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- FR801, Rennes, France